CLINICAL TRIAL: NCT04712175
Title: Validation Diagnostique de la détection Rapide du Virus SARS-CoV-2 Dans Des échantillons Salivaires Par spectrométrie de Masse
Brief Title: Diagnostic Validation of Rapid Detection of the COVID-19 Causative Virus (SARS-CoV-2) in Saliva Samples by Mass Spectrometry
Acronym: SALICOV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Technological Innovations for Detection and Diagnosis Laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: LOCAL-COVID/2020/AS-01
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Anonymized saliva samples of patients with positive RT-PCR results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SARS-CoV-2 infection
  Interventions: Diagnostic Test: Nasopharyngeal sampling; Diagnostic Test: Saliva sampling
- Patients without SARS-CoV-2 infection
  Interventions: Diagnostic Test: Nasopharyngeal sampling; Diagnostic Test: Saliva sampling

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal sampling — Swabs will be taken of nasopharyngeal samples for RT-PCR
Diagnostic Test: Saliva sampling — A 10ml saliva sample will collected in a sterile 60ml bottle for mass spectrometry and RT-PCR

SUMMARY:
In order to control the COVID-19 pandemic, a policy for the diagnosis and screening of people likely to be infected with SARS-CoV-2 has been established The reference diagnostic test is RT-PCR on nasopharyngeal swab. Nasopharyngeal swabbing requires training, generates a risk of aerosolization and therefore viral transmission to the operator, and is unpleasant or even painful for the patient. RT-PCR is efficient, but time-consuming. It is therefore necessary to consider techniques that are less subject to difficulties of production and sampling, and less time-consuming. Tandem mass spectrometry on saliva samples is a promising option. A combined "mass spectrometry/saliva test" should provide faster results.

ELIGIBILITY:
Inclusion Criteria:

* The patient must not have opposed their inclusion in the study
* Patient presenting to the Walk-in Center for Emerging Biological Risks for SARS-CoV-2 screening by nasopharyngeal swab OR hospitalized in the Infectious and Tropical Diseases Department for severe SARS-CoV-2 infection, diagnosed by RT-PCR on nasopharyngeal sample, taken at Nîmes University Hospital, in the previous 24 hours.

Exclusion Criteria:

* Patient already included in the study
* The subject is in a period of exclusion determined by a previous study
* It is impossible to give the subject clear information
* The patient is under safeguard of justice or state guardianship
* Patient unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the Walk-in Center for Emerging Biological Risks of the Nîmes University Hospital for screening for SARS-CoV-2 infection or who are hospitalized at the Infectious and Tropical Diseases Department for severe infection with SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 on nasopharyngeal samples (gold standard) | Day 0
  RT-PCR
Detection of SARS-CoV-2 on a saliva samples by mass spectrometry | Day 0
  tandem mass spectrometry test

SECONDARY OUTCOMES:
Detection of SARS-CoV-2 on saliva samples via RT-PCR | Day 0
  RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sotto, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Background] Gouveia D, Miotello G, Gallais F, Gaillard JC, Debroas S, Bellanger L, Lavigne JP, Sotto A, Grenga L, Pible O, Armengaud J. Proteotyping SARS-CoV-2 Virus from Nasopharyngeal Swabs: A Proof-of-Concept Focused on a 3 Min Mass Spectrometry Window. J Proteome Res. 2020 Nov 6;19(11):4407-4416. doi: 10.1021/acs.jproteome.0c00535. Epub 2020 Aug 5. PMID 32697082